CLINICAL TRIAL: NCT02096926
Title: Methodological Validation of Ibuprofen Verses Placebo for Post Operative Pain After Third Molar Extraction Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lotus Clinical Research, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCR-DEN-01C
Record Dates: First submitted 2014-03-24; First posted 2014-03-26 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Dental Pain
Keywords: Third Molar Extraction
MeSH Terms: conditions — Toothache | interventions — Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo
- Ibuprofen (Active Comparator): 400 mg PO
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: Ibuprofen — 400 mg PO
  Arms: Ibuprofen

SUMMARY:
This is a single center placebo controlled, prospective, randomized study on healthy adults undergoing third molar surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who provide written informed consent prior to enrollment
* Male or female and 18 to 40 years of age
* Patients who are scheduled to undergo elective ipsilateral two (2) third molar extraction surgery under local anesthesia The mandibular third molar must involve full or partial bony impaction confirmed by radiographic evidence
* Female subjects are eligible only if all of the following apply

  * Not pregnant (subjects of child bearing potential must have a negative urine beta human chorionic gonadotropin (β-hCG) pregnancy test before surgery)
  * Not lactating
  * Not planning to become pregnant within the duration of the study
* Patients who are willing and capable of understanding and cooperating with the requirements of the study
* Patients able to understand and communicate in English

Exclusion Criteria:

* Patients who have participated in a Lotus Clinical Research placebo response and pain scale education training program
* Patients with a medical condition that, in the Investigator's opinion, could adversely impact the patient's participation, safety, or conduct of the study such as but not limited to a history of severe renal or hepatic impairment, severe active hepatic disease, other acute or chronic pain conditions, or any other clinically significant medical condition
* Patients who have a known history of intolerance, severe allergy or hypersensitivity to Ibuprofen, opioid analgesics, Lidocaine, or acetaminophen (APAP)
* Patients who have abused any prescription medication or alcohol within two years before the start of the study
* Patients who have surgical complications that could compromise safety of the subject or confound the results of the study
* The subject is taking any corticosteroid chronically (except for an inhaled steroid for pulmonary disease) or has taken systemic corticosteroids within 4 weeks of the proposed date of surgery
* The subject is taking central nervous system (CNS) active drugs such as benzodiazepines, tricyclic antidepressants, selective serotonin reuptake inhibitors (SSRIs) or serotonin norepinephrine reuptake inhibitors (SNRIs) for pain. These drugs are permitted for non-pain indications throughout the study, if the dose has been stable for at least 30 days
* The subject has used acetylsalicylic acid, acetaminophen or nonsteroidal antiinflammatory drug (NSAIDs) within 5 half-lives prior to the planned day of the surgery
* The subject is taking an antihypertensive agent(s) or a diabetic regimen at a dose that has not been stable for at least 28 days.
* Patients who have a history of seizures, or are currently taking anticonvulsants
* Patients who have dysphagia and/or cannot swallow study medication whole
* Patient who is unable to adequately communicate with study staff, properly give informed consent, or otherwise comply with study procedures
* Patient who has participated in another clinical trial of an investigational drug or device within 30 days of screening visit or is schedule to receive an investigational product while participating in the study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Sum of pain intensity difference (SPID)6 | 6 hours

SECONDARY OUTCOMES:
Sum of pain intensity difference (SPID) 3 | 3 hour

OTHER OUTCOMES:
Total Pain Relief (TOTPAR) 6 | 6 hours
Patient Global Assessment | 6 hours post study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Singla, DO, Principal Investigator — Lotus Clinical Research, LLC
Locations (1):
- Lotus Clinical Research, LLC, Pasadena, California, United States